CLINICAL TRIAL: NCT05254145
Title: Insight of Joint Microbiome From Different Knee Conditions.
Brief Title: Joint Microbiome Study for the Knee
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: JPAR22D.042
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis; PJI
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A: This group will include participants without an arthritic knee. These participants will be recruited from the Orthopedic Sports Medicine consultation
  Interventions: Diagnostic Test: Next Generation Sequencing
- Group B: This group will include participants undergoing primary knee arthroplasty (KA).
  Interventions: Diagnostic Test: Next Generation Sequencing
- Group C: This group will include participants undergoing a surgical procedure whose opposite knee has no history of arthritis
  Interventions: Diagnostic Test: Next Generation Sequencing
- Group D: This group will include participants undergoing knee revision surgery with no suspicion of infection (aseptic knee revision replacement)
  Interventions: Diagnostic Test: Next Generation Sequencing
- Group E: This group will include participants undergoing knee revision with a known infection (septic knee revision replacements)
  Interventions: Diagnostic Test: Next Generation Sequencing

INTERVENTIONS:
Diagnostic Test: Next Generation Sequencing — During the participants surgical procedure, a total of 3 ml of synovial fluid (joint fluid collected from the knee) will be collected per joint. Upon collection, the samples will be deidentified, stored on ice and shipped with a study ID number to MicroGenDx for Next Generation Sequencing.

SUMMARY:
Prosthetic joint infection (PJI) is a devastating complication following arthroplasty. An utmost effort has been done to clarify risk factors and microbiology of PJI. We now know the most frequent infecting microorganisms are members of the skin microbiome. These microorganisms are thought to get into the joint and infect the prosthesis during the peri-operative and/or post-operative period. Nevertheless, recent studies have suggested, bacteria may be present in the joint even before the first incision, suggesting the existence of a joint microbiome. Therefore, we aimed to determine the bacterial composition from different knee conditions.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years or older who give verbal and written informed consent for the retrieval of experimental samples and data collection.
* Group A: Subjects with lack of Osteoarthritis (OA) evidence, invasive examinations, minor procedures, cartilage damage, and/or synovitis in joints.
* Group B: Patients undergoing primary knee arthroplasty (partial or total).
* Group C: Contralateral non-affected (native) joint without knee arthroplasty, history of septic arthritis (SA), invasive examinations and/or minor procedures.
* Group D: Patients undergoing aseptic knee revision surgery.
* Group E: Patients undergoing septic knee revision surgery

Exclusion Criteria:

* Withdrawal of informed consent, suspicion of PJI, surgical site infection (SSI) or septic arthritis (SA) before samples retrieval, use of antibiotics within 4 weeks before collecting the samples (not including perioperative antimicrobial prophylaxis), inflammatory arthritis, systemic rheumatic disorder, high risk of infection.
* Group A: History and/or suspicion before/at samples retrieval of SA in native joint.
* Group B: History and/or suspicion before/at samples retrieval of SSI or SA in the affected joint.
* Group C: No additional criterion.
* Group D: History and/or suspicion before/at samples retrieval of PJI, SSI, SA in the affected joint
* Group E: No additional criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited preoperatively during their elective procedure scheduling visit (diagnostic/treatment algorithm for group A or surgery for groups B-E, accordingly). Patients presenting for Orthopedic Sports Medicine consultation (group A), with end-stage knee osteoarthritis who are candidates for TKA (group B/C), patients with a TKA who require an aseptic knee revision surgery (group C/D), or those patients complicated by PJI (group E), and who agree to participate in the study will undergo the informed consent process
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-20 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Determine the microbiome (bacterial composition) of the knee joint | 3 days
  Joint fluid taken from the operative knee during surgery will be analyzed using next generation sequencing (NGS).

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States